CLINICAL TRIAL: NCT00753883
Title: A Randomized, Open-Labeled, Parallel Group Comparison Study to Evaluate the Efficacy, Safety of Ezetimibe Alone Versus Statin in the Treatment of Hypercholesterolemia
Brief Title: Ezetrol Post-Marketing Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008_024; MK0653-154
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Simvastatin; Ezetimibe

ARMS (2):
- 1 (Active Comparator): simvastatin 20 mg/qd for 8 weeks, and then add on ezetrol 10mg (if ldl-c . 160mg/dl) for another 8 weeks.
  Interventions: Drug: simvastatin; Drug: Ezetimibe
- 2 (Active Comparator): ezetrol 10 mg/qd for 8 weeks, and then add on simvastatin 20 mg qd (if ldl-c . 160mg/dl) for another 8 weeks
  Interventions: Drug: simvastatin; Drug: Ezetimibe

INTERVENTIONS:
Drug: simvastatin — simvastatin 20 mg/QD for 6 Weeks.
  Other Names: MK0733; Zocor®
Drug: Ezetimibe — Ezetimibe 10 mg/QD for 8 weeks.
  Other Names: Ezetrol; Zetia; MK0653

SUMMARY:
To compare the lipid lowering efficacy of adding ezetimibe to statin vs. statin alone.

ELIGIBILITY:
Inclusion Criteria:

* Men Or Women Older Than 20 And Younger Than 80 Years Of Age
* Willing To Follow An Ncep Therapeutic Lifestyle Changes (TLC) Or Similar Cholesterol-Lowering Diet For The Duration Of The Study
* Female Patients Receiving Hormone Therapy (Including Hormone Replacement Therapy, And Estrogen Antagonist/Agonist, Or Oral Contraceptives) If Maintained On A Stable Dose And Regimen For At Least 8 Weeks Prior To Visit 1 And If Willing To Continue The Same Regimen Throughout The Study
* Patient With Total Cholesterol Equal Or Greater Than 240 Mg/Dl Or Ldl-C Equal Or Greater Than 160 Mg/Dl For Primary (Heterozygous Familial And Non-Familial) Hypercholesterolemia And/Or Ldl-C Equal Or Greater Than 130 Mg/Dl For Secondary Hypercholesterolemia With Identifiable Risk Factors
* Patient Is Able To Discontinue Any Lipid Lowering Drugs For 6-8 Weeks Wash-Out Period (6 Week For Statin And 8 Week For Fibrate)
* Triglyceride (Tg) Concentrations Equal Or Less Than 400 Mg/Dl
* Liver Transaminases (Alt, Ast) Equal Or Less Than 1.5x Uln With No Active Liver Disease And Equal Or Less Than 1.5x Uln At Visit 2

Exclusion Criteria:

* Women Who Are Pregnant Or Lactating
* History Of Mental Instability, Drug/Alcohol Abuse Within The Past 5 Years, Or Major Psychiatric Illness Not Adequately Controlled And Stable On Pharmacotherapy
* Patients Who Have Been Treated With Any Other Investigational Drug Within 3 Months Of Visit 1
* Patients Previously Randomized To A Study With Ezetimibe
* Active Liver Disease Or Impaired Liver Function Tests (Alt, Ast > 1.5xuln)
* Impaired Renal Function ( Serum Creatinine Equal Or Greater Than 1.5 Mg/Dl Or Urine Protein Equal Or Greater Than 100 Mg/L) Or Nephritic Syndrome At Visit 1
* Unstable Angina
* Myocardial Infarction, Coronary Bypass Surgery Or Angioplasty Within The Previous Three Months Of Visit 1
* Uncontrolled Cardiac Arrhythmias
* Uncontrolled Hypertension (Treated Or Untreated) With Systolic Blood Pressure > 160 Mmhg Or Diastolic > 100 Mmhg At Visit 1
* Poorly Controlled Diabetes Mellitus Patient. (Hba1c>8.0%). If The Patient Treated With Md, No Any Dm Medication Will Be Change During The Study Period)
* Uncontrolled Endocrine Or Metabolic Disease Known To Influence Serum Lipids Or Lipoprotein, E.G. Hyperthyroidism (Tsh > 5.5 (Iu/Ml). However, Patients Who Are On A Stable Therapy Of Thyroid Replacement Therapy For At Least 6 Weeks Are Eligible For Enrollment
* Patients Hypersensitive To Hmg-Coa Reductase Inhibitors Or Ezetimibe
* Patient Who Is Unable To Give Informed Consent (The Patient With A Legal Representative To Sign The Informed Consent Is Eligible To Participate The Study.)
* Any Condition Or Situation Which, In The Opinion Of The Investigator, Might Pose A Risk To The Patient Or Confound The Results Of The Study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The change in lipid profiles after study drug treatment. | After 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC